CLINICAL TRIAL: NCT01682343
Title: Effect of High-calcium Intake on Appetite, Insulinemia and Incretins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD Student, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 32AN2
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Nutritional and Metabolic Diseases
MeSH Terms: conditions — Nutritional and Metabolic Diseases | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Breakfast consisting of milk-based porridge with a normal calcium content.
- High-Calcium (Experimental): As control, but with a high-calcium content.
  Interventions: Dietary Supplement: Calcium

INTERVENTIONS:
Dietary Supplement: Calcium — Milk-calcium supplement
  Arms: High-Calcium

SUMMARY:
The purpose of this study is to investigate the appetite, insulin and incretin hormone responses to a high-calcium meal.

DETAILED DESCRIPTION:
Participants will be provided with control and high-calcium meals. Insulin, appetite, glucagon-like peptide-1 and glucose-dependent insulinotropic peptide responses will be assessed, along with rates of substrate oxidation.

ELIGIBILITY:
Inclusion Criteria:

* recreationally active
* male

Exclusion Criteria:

* food intolerances/allergies

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Subjective appetite ratings | 3 hour
  Subjective ratings of appetite assessed by visual analogue scales.

SECONDARY OUTCOMES:
Serum insulin concentration | 2 hour
  2 hour area under the curve for serum insulin following breakfast consumption
Plasma glucose-dependent insulinotropic peptide concentration | 2 hour
  2 hour area under the curve for plasma glucose-dependent insulinotropic peptide following breakfast consumption
Plasma glucagon-like peptide-1 concentration | 2 hour
  2 hour area under the curve for plasma glucagon-like peptide-1 following breakfast consumption

OTHER OUTCOMES:
Total fat oxidised during 60 min of exercise (g) | 1 hour
  Assessed by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Javier T Gonzalez, MRes, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne on Wear, United Kingdom